CLINICAL TRIAL: NCT00328510
Title: A Randomized Trial Comparing Two Forms of Immobilization of the Head for Fractioned Stereotactic Radiotherapy
Brief Title: Comparing Two Forms of Head Immobilization for Stereotactic Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04U.534; 2004-72 (Other: CCRRC)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Patients Receiving Fractionated Stereotactic Radiotherapy; for Brain Tumors
Keywords: Stereotactic radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTC Frame (Experimental): Participant undergoes SRT using a GTC frame to immobilize the participant's heading during radiation therapy
  Interventions: Device: GTC frame; Radiation: Stereotactic radiation therapy
- BrainLab thermoplastic mask (Experimental): Participant undergoes SRT using the BrainLab thermoplastic mask to immobilize the participant's head during radiation therapy
  Interventions: Device: Thermoplastic facemask; Radiation: Stereotactic radiation therapy

INTERVENTIONS:
Device: GTC frame
  Arms: GTC Frame
Device: Thermoplastic facemask
  Arms: BrainLab thermoplastic mask
Radiation: Stereotactic radiation therapy
  Other Names: SRT

SUMMARY:
Fractionated stereotactic radiotherapy (SRT) requires extremely precise and reproducible immobilization of the patient's head. This randomized study compares the efficacy of two commonly used forms of immobilization used for SRT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1) To compare the efficacy of two commonly used, generally accepted forms of immobilization for the treatment of lesions in the head with fractionated stereotactic radiotherapy. Specifically, this study will use the ExacTRAC kilovoltage imaging system to assess positioning accuracy for these two systems.

OUTLINE:

Two routinely used methods of immobilization, which differ in their approach to reproduce head position from day-to-day are the Gill-Thomas-Cosman (GTC)frame and the BrainLab thermoplastic mask. The GTC frame fixates on the patient upper detention and thus us in direct mechanical contact with the cranium. The BrainLab mask is a two-part masking system custom-fitted to the front and back of the participant's head. After patients sign an IRB-approved informed consent form, eligible participants are either randomized to either the GTC frame or the mask for their course of SRT. Participants are treated as per standard procedure; however, prior to each treatment, a set of digital kV images (ExacTrac, BrainLabAB, Germany) is taken. These images are fused with reference digitally constructed radiographs obtained from treatment planning CT to yield lateral, longitudinal, and vertical deviations of isocenter and head rotations about respective axes. The primary endpoint of the study is to compare the two systems with respect to mean and standard deviations (SDs) using the distance to isocenter measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for fractionated stereotactic radiotherapy

Exclusion Criteria:

* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Shiu A, Parker B, Ye JS, Lii J. An integrated treatment delivery system for CSRS and CSRT and clinical applications. J Appl Clin Med Phys. 2003 Autumn;4(4):261-73. doi: 10.1120/jacmp.v4i4.2496. PMID 14604415
- [Background] Burton KE, Thomas SJ, Whitney D, Routsis DS, Benson RJ, Burnet NG. Accuracy of a relocatable stereotactic radiotherapy head frame evaluated by use of a depth helmet. Clin Oncol (R Coll Radiol). 2002 Feb;14(1):31-9. doi: 10.1053/clon.2001.0001. PMID 11898783
- [Background] Lopatta E, Liesenfeld SM, Bank P, Wurm R, Gunther R, Wiezorek T, Wendt TG. [Improved patient repositioning accuracy by integrating an additional jaw fixation into a high precision face mask system in stereotactic radiotherapy of the head]. Strahlenther Onkol. 2003 Aug;179(8):571-5. doi: 10.1007/s00066-003-0941-3. German. PMID 14509957
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.kimmelcancercenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GTC Frame | BrainLab Thermoplastic Mask
Started | 42 | 41
Completed | 32 | 37
Not Completed | 10 | 4
Not completed — Gag disorder, could not use frame | 4 | 0
Not completed — Dentition problems, could not use frame | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Severe kyphosis, could not use mask | 0 | 1
Not completed — Treatment changed to a single fraction | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GTC Frame | BrainLab Thermoplastic Mask | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (14.93) | 56.94 (14.07) | 56.18 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Distance From Ideal to Center of GTC Frame and BrainLab Thermoplastic Mask With Respect to Average and Variability
Description: This study uses the ExacTRAC imaging system to assess positioning of frame or mask during SRT. Images yield lateral, longitudinal, and vertical deviations of the isocenter as well as head rotations about respective axes.
Time Frame: Measurements taken during SRT
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Measurements
Arm/Group | GTC Frame | BrainLab Thermoplastic Mask
Number analyzed (Participants) | 32 | 37
Number analyzed (Measurements) | 714 | 782
millimeters | 2.00 (1.04) | 3.17 (1.95)

ADVERSE EVENTS:
Arm/Group | GTC Frame | BrainLab Thermoplastic Mask
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/37
Other Adverse Events (participants affected / at risk) | 0/32 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes